CLINICAL TRIAL: NCT00872105
Title: A Multicentre, Randomized Trial of Conservative Treatment Versus Operative Plate Fixation for Acute, Displaced Fractures of the Distal Clavicle
Brief Title: Conservative Treatment Versus Operative Plate Fixation for Acute, Displaced Fractures of the Distal Clavicle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Fraser Health (Other); University of British Columbia (Other); London Health Sciences Centre (Other); University of Calgary (Other); Nova Scotia Health Authority (Other); Winnipeg Regional Health Authority (Other); McGill University Health Centre/Research Institute of the McGill University Health Centre (Other); The Ottawa Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Distal Clavicle Study
Record Dates: First submitted 2009-03-30; First posted 2009-03-31 (Estimated); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Clavicle Fracture; Fractures
Keywords: clavicle; fractures; distal
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Non-operative treatment (Other): The first treatment strategy will involve conservative (nonoperative) management of the clavicle fracture.
  Interventions: Procedure: Non-operative Treatment
- Operative treatment (Active Comparator): The second treatment strategy will involve operative fixation (i.e. ORIF) of the fracture with a plate and screws.
  Interventions: Procedure: Operative Treatment

INTERVENTIONS:
Procedure: Non-operative Treatment — Standard protocol for conservative treatment will consist of the implementation of a sling, for clavicular support and patient comfort. Pendulum or gentle Range of Motion (ROM) shoulder exercises may be implemented at any time as dictated by the attending surgeon.
  Arms: Non-operative treatment
Procedure: Operative Treatment — The operating surgeon will determine the positioning of the patient for surgery. ORIF of the distal clavicle fracture will be carried out as follows:
  Anatomic reduction of the fracture Definitive fixation with a contoured clavicle plate and screws; a AO hook plate; a 3.5 LCDC, reconstruction, or compression plate is acceptable; a 1/3 tubular plate is not acceptable Use of bone graft is optional (iliac crest bone autograft)
  Arms: Operative treatment

SUMMARY:
This is a multicentre randomized clinical trial prospectively comparing operative treatment versus conservative (nonoperative) care in the management of displaced distal (Type II) clavicle fractures.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 16 to 60 years of age
* Completely displaced (no cortical contact), closed fracture of the distal 3rd of the clavicle (Type II) confirmed by radiograph
* Fractures within 28 days post injury
* Provision of informed consent

Exclusion Criteria:

* Pathological fractures
* Non-displaced (cortical contact) distal clavicle fractures
* Open clavicle fractures
* Presence of vascular injury
* Fractures more than 28 days post-injury
* Limited life expectancy due to significant medical co-morbidity
* Medical contraindication to surgery
* Inability to comply with rehabilitation or form completion
* Likely problems, in the judgement of the investigators, with maintaining follow-up (i.e. patients with no fixed address, patients not mentally competent to give consent, etc.)

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 59 (Actual)
Dates: Start 2009-03; Primary Completion 2018-12 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
The primary outcome measurement will be patient DASH (Disabilities of the Arm, Shoulder and Hand Instrument) scores. The DASH is a patient-oriented, limb-specific, functional measurement questionnaire. | 2 years

SECONDARY OUTCOMES:
The secondary outcome measurement patients' functional shoulder scores as defined by Constant's Shoulder Score (i.e. pain, activities of daily living, range of motion and power). | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy A Hall, MD, FRCS(C), Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada